CLINICAL TRIAL: NCT01197495
Title: Safety and Effectiveness of Juvederm(R) Ultra XC Injectable Gel for Lip Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: JULIDO-002
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2016-06-07 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Juvederm(R) Ultra XC Injectable Gel
  Interventions: Device: hyaluronic acid gel
- Control (Experimental): No treatment for 3 months followed by Juvederm(R) Ultra XC Injectable Gel at Month 3.
  Interventions: Device: hyaluronic acid gel

INTERVENTIONS:
Device: hyaluronic acid gel — Dosage per Investigator's discretion to obtain lip treatment gel; 1 touch-up treatment is allowed 14 to 30 days after initial treatment. Repeat treatment occurs at month 12. Subjects in the control group start with treatment at month 3. Maximum total volume per subject is 4.8 mL for initial and touch-up treatment combined.
  Other Names: Juvederm(R) Ultra XC Injectable Gel

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of Juvederm(R) Ultra XC Injectable Gel for lip augmentation

DETAILED DESCRIPTION:
All subjects were randomized to either the treatment group, Juvederm(R) Ultra XC Injectable Gel, or to the control group (no treatment). At month 3, subjects in the control group crossed over to the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Desire augmentation of his/her lips
* Have a pre-treatment score of Minimal or Mild

Exclusion Criteria:

* Have lip tattoos, facial hair or scars that would interfere with visualization of the lips and perioral area for the effectiveness assessments
* Have dentures or any device covering all or part of the upper palate, and/or severe malocclusion, dentofacial or maxillofacial deformities, or significant asymmetry of the lips and perioral area, as judged by the Treating Investigator
* Have undergone oral surgery or other dental procedures (e.g., tooth extraction, orthodontia, or implantation) within 30 days prior to enrollment or be planning to undergo any of these procedures during the study
* Have ever undergone facial plastic surgery or received semi-permanent fillers or permanent facial implants (e.g., calcium hydroxylapatite, L-polylactic acid, PMMA, silicone, ePTFE) anywhere in the face or neck, or be planning to be implanted with any of these products at any time during the study
* Have undergone temporary dermal filler treatment within 24 months prior to study entry or be planning to undergo any of these procedures at any time during the study
* Have undergone cosmetic facial procedures, e.g., resurfacing (laser photomodulation, intense pulsed light, radio frequency, dermabrasion, chemical peel, or other ablative or non-ablative procedures) or mesotherapy anywhere in the face or neck, or BOTOX® Cosmetic injections in the lower face (below the orbital rim), within 6 months prior to entry in the study or be planning to undergo any of these procedures at any time during the study
* Begin use of any new over-the-counter or prescription, oral or topical, anti-wrinkle products for the lips or around the mouth within 3 months (90 days) prior to enrollment or be planning to begin use of such products at any time during the study [NOTE: use of sunscreens and continued therapy with some cosmeceuticals (e.g., alpha hydroxy acids, glycolic acids, retinol, or retinoic acids) is allowed if the regimen was established ≥ 3months (90 days) prior to enrollment and the regimen remains unchanged during the study
* Have a history of anaphylaxis, multiple severe allergies, atopy, allergy to lidocaine, hyaluronic acid products or Streptococcal protein, or be planning to undergo desensitization therapy during the term of the study
* Have an active inflammation, infection, cancerous or pre-cancerous lesion, or unhealed wound in the mouth area
* Be on an ongoing regimen of anti-coagulation therapy (e.g., warfarin) or have taken NSAIDS (e.g., aspirin, ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with garlic or gingko) within 10 days of undergoing study device injections [Study device injections may be delayed as necessary to accommodate this 10-day washout period.]
* Be pregnant, lactating, or planning to become pregnant at any time during the study
* Have received investigational product within 30 days prior to study enrollment or be planning to participate in another investigation during the course of this study
* Be an employee (or immediate relative of an employee) of the Treating Investigator, Evaluating Investigator, Sponsor or representative of the Sponsor
* Have a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2014-06-19 (Actual); Study Completion 2015-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nashville, Tennessee, United States

REFERENCES:
- [Background] Dayan S, Bruce S, Kilmer S, Dover JS, Downie JB, Taylor SC, Skorupa A, Murphy DK. Safety and Effectiveness of the Hyaluronic Acid Filler, HYC-24L, for Lip and Perioral Augmentation. Dermatol Surg. 2015 Dec;41 Suppl 1:S293-301. doi: 10.1097/DSS.0000000000000540. PMID 26618456

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The modified intent-to-treat (mITT) population is presented and includes all treated subjects.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 157 | 56
Completed | 144 | 49
Not Completed | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 157 | 56 | 213
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (11.46) | 49.2 (9.72) | 48.8 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 54 | 204
  Male | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With ≥1-Point Improvement on the Investigator Assessed 5-point Lip Fullness Scale 2 (LFS2)
Description: Overall lip fullness is assessed by the blinded Evaluating Investigator compared to baseline using the 5-point LFS2. Scores range from 1=minimal improvement to 5=very marked improvement.
Time Frame: Baseline, Month 3
Population: Modified Intent-to-Treat: all treated subjects with data at the designated time point
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Treatment | Control
Number analyzed (Participants) | 139 | 46
Percentage of Subjects | 79.1 [71.43 to 85.56] | 26.1 [14.27 to 41.13]

2. Secondary Outcome: Percentage of Subjects With ≥1-Point Improvement on the Perioral Line (POL) Severity Scale
Description: Subject's upper lip perioral lines are assessed compared to baseline using the 4-point validated POL Severity Scale. Scores range from 0=None (best) to 3=Severe (worst).
Time Frame: Baseline, Month 3
Population: Subjects treated for POL at the designated time points
Measure: Number; unit: Percentage of Subjects
Arm/Group | Treatment
Number analyzed (Participants) | 61
Percentage of Subjects | 47.5

3. Secondary Outcome: Percentage of Oral Commissures With ≥1-Point Improvement on the Oral Commissures Severity (OCS) Scale
Description: Subject's right and left oral commissures are assessed compared to baseline using the validated OCS Scale. Scores range from 0=none (best) to 3=severe (worst).
Time Frame: Baseline, Month 3
Population: Subjects treated for OCS at the designated time points
Measure: Number; unit: Percentage of Oral Commissures
Units Other Than Participants: Oral Commissures
Arm/Group | Treatment
Number analyzed (Participants) | 157
Number analyzed (Oral Commissures) | 241
Percentage of Oral Commissures | 47.3

4. Secondary Outcome: Percentage of Subjects Achieving Their Personal Treatment Goal of Overall Lip Fullness
Description: Subjects assessed their personal treatment goal of overall lip fullness as 'achieved' or 'not achieved.'
Time Frame: Baseline, Month 3
Population: Treated subjects in the Treatment group
Measure: Number; unit: Percentage of Subjects
Arm/Group | Treatment
Number analyzed (Participants) | 137
Percentage of Subjects | 81.8

5. Secondary Outcome: Duration Effect of Treatment on Lip Fullness
Description: Duration of treatment effect on lip fullness is assessed by the blinded Evaluating Investigator as ≥1-point Improvement from baseline in overall lip fullness of the eligible lip at each visit.
Time Frame: Month 1, Month 3, Month 6, Month 7.5, Month 9, Month 10.5, Month 12
Population: Modified Intent-to-Treat: all treated subjects with data at the designated time point
Measure: Number (95% Confidence Interval); unit: % of Pts Retaining ≥1-point Improvement
Arm/Group | Treatment | Control
Number analyzed (Participants) | 142 | 48
% of Pts Retaining ≥1-point Improvement
  Month 1 | 93.5 [89.53 to 97.38] | 98.0 [94.00 to 100.0]
  Month 3 (N=114, 37) | 77.5 [70.78 to 84.13] | 77.3 [65.42 to 89.08]
  Month 6 (N=99, 35) | 69.1 [61.64 to 76.54] | 74.8 [62.34 to 87.18]
  Month 7.5 (N=89, 29) | 64.4 [56.51 to 72.20] | 63.9 [49.37 to 78.36]
  Month 9 (N=75, 24) | 54.1 [45.58 to 62.54] | 55.4 [39.97 to 70.82]
  Month 10.5 (N=69, 19) | 48.9 [40.29 to 57.53] | 45.8 [29.64 to 61.92]
  Month 12 (N=51, 8) | 45.1 [36.32 to 53.78] | 36.6 [16.02 to 57.23]

ADVERSE EVENTS:
Description: 208 subjects includes subjects who received initial treatment in both groups (157 in the treatment group and 51 in the control group).
  114 subjects includes subjects who had repeat treatment from both treatment groups.
Groups:
- Onset Prior to Repeat Treatment; Onset After Repeat Treatment: Juvederm(R) Ultra XC Injectable Gel
Arm/Group | Onset Prior to Repeat Treatment | Onset After Repeat Treatment
Serious Adverse Events (participants affected / at risk) | 4/208 | 2/114
Other Adverse Events (participants affected / at risk) | 63/208 | 28/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Onset Prior to Repeat Treatment (N=208) | Onset After Repeat Treatment (N=114)
Development Hip Dysplasia (Congenital, familial and genetic disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Premature Baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Onset Prior to Repeat Treatment (N=208) | Onset After Repeat Treatment (N=114)
Injection Site Mass (General disorders) | 33 | 11
Injection Site Induration (General disorders) | 21 | 11
Injection Site Pain (General disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.